CLINICAL TRIAL: NCT05640674
Title: A Randomized Controlled Trial of Opioid vs Non-Opioid Postoperative Pain Management in Children With Supracondylar Humerus Fractures
Brief Title: Post-operative Pain Management in Children With Supracondylar Humerus Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After reviewing our enrollment numbers and feasibility, we have decided to close the study due to low enrollment.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Scott Rosenfeld, Associate Professor of Orthopaedic Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 52475
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Supracondylar Humerus Fracture
MeSH Terms: interventions — Ibuprofen; oxycodone-acetaminophen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid Pain Management (Active Comparator): Ibuprofen (liquid, 10mg/kg/dose every 6 hours) will be the first line pain medication and Hydrocodone/Acetaminophen (liquid, 0.135mg Hydrocodone/kg/dose every 6 hours) will be used as needed for breakthrough pain.
  Interventions: Drug: Ibuprofen; Drug: Hydrocodone/acetaminophen
- Non-Opioid Pain Management (Experimental): Ibuprofen (liquid, 10mg/kg/dose every 6 hours) will be the first line pain medication and Acetaminophen (liquid, 15mg/kg/dose every 6 hours) will be used as needed for breakthrough pain.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — Non-opioid
  Other Names: Motrin, Advil
Drug: Hydrocodone/acetaminophen — Opioid
  Other Names: Hycet
  Arms: Opioid Pain Management
Drug: Acetaminophen — Non-opioid
  Other Names: Tylenol
  Arms: Non-Opioid Pain Management

SUMMARY:
There are two common and concurrently used strategies for pain management following surgical treatment of supracondylar humerus (elbow) fractures in children: opioids vs over the counter pain medications. The purpose of this study is to determine if ibuprofen and acetaminophen can provide similar or better pain relief compared to ibuprofen and hydrocodone/acetaminophen (also known as Hycet) for this population of children after they have been discharged. If over the counter medications can provide adequate pain relief, then fewer opioid prescriptions would be necessary. This reduces early opioid exposure and decreases unnecessary opioids in circulation.

DETAILED DESCRIPTION:
Prior to surgery, participants will be randomly assigned to a group that will determine whether they are prescribed an opioid vs non-opioid pain management plan at discharge. Each participants' parent or guardian will be given a journal to keep track of their child's pain severity and the pain medications taken. The journal will updated daily until participants no longer require pain medication. Participants will follow up with their surgeon per usual at their post-operative visits.

ELIGIBILITY:
Inclusion Criteria:

* Closed, Gartland type III supracondylar humerus fracture
* Fractures treated with closed reduction and percutaneous pinning (CRPP)
* Patients expected to follow up at Texas Children's Hospital
* Patients/guardians must speak English or Spanish

Exclusion Criteria:

* Fractures associated with open skin wounds, polytrauma, neurologic deficit, or vascular deficit
* Patients who have impaired ability to report pain severity such as intellectual delay.
* Patients who have a problem with bone healing such as osteogenesis imperfecta.
* Patients who are unable to take the standard dose of acetaminophen, ibuprofen, or hydrocodone (allergy, severe kidney disease, etc).
* Patients who are on chronic NSAID or opioid medication prior to injury.
* Patients with injury from suspected non-accidental trauma.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rosenfeld, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Texas Children's Hospital - Main Campus, Houston, Texas
  - Texas Children's Hospital - West Campus, Houston, Texas
  - Texas Children's Hospital - Woodlands Campus, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid Pain Management | Non-Opioid Pain Management
Started | 14 | 15
Completed | 8 | 5
Not Completed | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Pain Management | Non-Opioid Pain Management | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.6 (2.2) | 6.4 (1.3) | 6.5 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 1 | 10 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 6 | 16
  Black | 1 | 1 | 2
  Hispanic | 3 | 7 | 10
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Daily Pain Scores on the FACES Scale
Description: A parent/guardian will ask participants to rate their pain severity using the Wong-Baker FACES scale, which ranges from 0 (no pain) to 10 (worst pain).
Time Frame: from discharge until pain medication is no longer required (assessed up to 3 weeks)
Population: Only 8 opioid and 5 non-opioid patients completed the pain journal, so they are the only patients who could be analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale/day
Arm/Group | Opioid Pain Management | Non-Opioid Pain Management
Number analyzed (Participants) | 8 | 5
scores on a scale/day | 2.7 (3.0) | 1.31 (1.9)

2. Secondary Outcome: Number of Days Pain Medication Required
Description: A parent/guardian will record the doses of pain medications given to the participant each day.
Time Frame: from discharge until pain medication is no longer required (assessed up to 3 weeks)
Population: Only 8 opioid and 5 non-opioid patients completed the pain journal, so they are the only patients who could be analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Opioid Pain Management | Non-Opioid Pain Management
Number analyzed (Participants) | 8 | 5
days | 12.5 (7.13) | 6.2 (2.49)

3. Secondary Outcome: Number of Pain Medication Doses Required Per Day
Description: A parent/guardian will record the doses of pain medications given to the participant each day.
Time Frame: from discharge until pain medication is no longer required (assessed up to 3 weeks)
Population: Only 8 opioid and 5 non-opioid patients completed the pain journal, so they are the only patients who could be analyzed.
Measure: Mean (Standard Deviation); unit: doses of medication/day
Arm/Group | Opioid Pain Management | Non-Opioid Pain Management
Number analyzed (Participants) | 8 | 5
doses of medication/day | 1.49 (0.5) | 1.42 (0.56)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 4 weeks
Arm/Group | Opioid Pain Management | Non-Opioid Pain Management
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

LIMITATIONS AND CAVEATS:
The study was terminated early due to insufficient enrollment, resulting in inadequate data to meaningfully assess the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT05640674/Prot_SAP_001.pdf